CLINICAL TRIAL: NCT00932945
Title: Monocentric Study, Phase III, for Safety Dermatological Evaluation: Acceptability With Gynaecological Follow up - Dermacyd PH_DESILSTY_FR (Lactic Acid).
Brief Title: Dermacyd PH_DESILSTY_FR (Lactic Acid) - Acceptability - Stay on Frutal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LACAC_L_04806
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Hygiene

ARMS (1):
- Dermacyd PH_DESILSTY_FR (Lactic Acid) (Experimental): Treatment duration: 21 consecutive days
  Interventions: Drug: LACTIC ACID(ND)

INTERVENTIONS:
Drug: LACTIC ACID(ND) — Treatment duration: 21 consecutive days

SUMMARY:
Primary Objective:

To prove the safety of the gynecological formulation in normal conditions of use.

ELIGIBILITY:
Exclusion criteria:

* Integral vaginal mucosa in the product analysis region
* Use the same category of cosmetics products
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time

Exclusion criteria:

* Use of Anti-inflammatory, immunossupression or antihistaminics drugs
* Allergic or atopic history to cosmetics products
* Cutaneous active disease (local and/or general) in the evaluated area
* Disease which can cause immunosuppresion, such as diabetes, HIV
* Endocrinology pathology such as thyroid gland, ovary and adrenal gland
* Intensive solar exposure until 15 days before evaluation
* Gynecological treatment until four weeks before the study
* Other reason considered by the investigator as a reason for not being included.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the absence of irritation and the good acceptability by using one specific scale which describes the intensity of the reaction. | From the treatment start up to the end of the study (treatment period 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil